CLINICAL TRIAL: NCT02705534
Title: Sustained Viral Response Rate in 50 Subjects With Cirrhosis Due to Hepatitis C, Genotype 1, Treated With 12 Weeks of Sofosbuvir, Ledipasvir and Ribavirin
Brief Title: Sofosbuvir, Ledipasvir, Ribavirin for Hepatitis C Cirrhotics, Genotype 1
Acronym: SL50
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Collaborators: Bakhtar Bioshimi Co (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 94-04-37-31023
Record Dates: First submitted 2016-03-07; First posted 2016-03-10 (Estimated); Last update posted 2018-04-30 (Actual); Status verified 2017-02

CONDITIONS: Hepatitis C; Cirrhosis
Keywords: Hepatitis C; Cirrhosis; Sofosbuvir; Ledipasvir; Ribavirin
MeSH Terms: conditions — Hepatitis C; Fibrosis | interventions — Sofosbuvir; ledipasvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Subjects will receive sofosbuvir, ledipasvir and ribavirin
  Interventions: Drug: Sofosbuvir; Drug: Ledipasvir; Drug: Ribavirin

INTERVENTIONS:
Drug: Sofosbuvir — 400 mg, included in a combination pill with 90 mg ledipasvir
  Other Names: SOF
Drug: Ledipasvir — 90 mg, included in a combination pill with 400 mg sofosbuvir
  Other Names: LDV
Drug: Ribavirin — 1000 mg/day if <75 kg, 1200 mg/day for >75 kg. Divided into two daily doses
  Other Names: RBV

SUMMARY:
The investigators will treat 50 patients with cirrhosis due to hepatitis C genotype 1, with sofosbuvir 400 mg daily, ledipasvir 90 mg daily and weight-based ribavirin (1000 mg/d if <75 kg, 1200 mg/d if >75 kg, divided in two daily doses) for 12 weeks and calculate the sustained viral response rate at 12 weeks.

DETAILED DESCRIPTION:
Cirrhosis due to Hepatitis C virus (HCV) presents a rather difficult treatment problem as many cannot tolerate interferon, the previous standard of care. The new direct acting antivirals have provided these patients with a new hope. One such combination is sofosbuvir (SOF) 400 mg and ledipasvir (LDV) 90 mg given once daily with or without weight-based ribavirin (RBV) for 12 or 24 weeks only for HCV genotype 1 patients. The current recommendation for cirrhotics (genotype 1) is SOF/LDV/RBV for 24 weeks but that recommendation is based on the lack of data for shorter periods. In order to evaluate the response rate to the combination of SOF/LDV/RBV the investigators decided to treat 50 HCV genotype 1 cirrhotics with this combination for 12 weeks. Patients with MELD score > 20 are excluded. The investigators will calculate the sustained viral response rate at 12 weeks (SVR12).

ELIGIBILITY:
Inclusion Criteria:

* Positive qualitative hepatitis C RNA polymerase chain reaction assay on two occasions at least 6 months apart

Exclusion Criteria:

* Renal failure [estimated glomerular filtration rate (eGFR) < 30 cc/min],
* Model or End stage Liver Disease (MELD) score > 20,
* Child's class C (score > 12),
* Heart rate < 50/min,
* Taking amiodarone

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
The sustained viral response rate | week 24 (12 weeks after end of treatment)
  Qualitative polymerase chain reaction assay for Hepatitis C RNA

SECONDARY OUTCOMES:
Adverse drug events | week 2, 4, 8, 12, 24
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Reza Malekzadeh, M.D., Study Chair — Tehran University of Medical Sciences
Locations (1):
- Shariati Hospital, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No